CLINICAL TRIAL: NCT03941951
Title: Quasi-experimental Intervention Study to Optimize the Use of New Antibiotics (Project NEW_SAFE)
Brief Title: Study to Optimize the Use of New Antibiotics
Acronym: NEW_SAFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FIS-TED-2019-01
Record Dates: First submitted 2019-04-04; First posted 2019-05-08 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Bacterial Infections; Fungal Infection
Keywords: Quasi-experimental study; Multidrug resistant bacteria; Antimicrobial stewardship; Ceftaroline; Tedizolid; Dalbavancin; Ceftazidime-avibactam; Ceftolozane-tazobactam; Isavuconazole
MeSH Terms: conditions — Bacterial Infections; Mycoses

STUDY DESIGN:
Intervention Model Description: The prescribers are assigned to receive the intervention if they have prescribed any of the antibiotics ceftaroline, tedizolid, dalbavancin, ceftazidime-avibactam, ceftolozane-tazobactam or isavuconazole from January 2010 to June 2021.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-intervention Cohort (No Intervention): Cohort of patients who have received either empirical or targeted treatment with ceftaroline, tedizolid, dalbavancin, ceftazidime-avibactam, ceftolozane-tazobactam or isavuconazole from January 2016 to December 2019 will be included.
- Intervention cohort (Other): Cohort of patients with complex infections treated with ceftaroline, tedizolid, dalbavancin, ceftazidime-avibactam, ceftolozane-tazobactam or isavuconazole from January 2010 to June 2021.
  Interventions: Behavioral: Non-impositive Program for Optimizing the Use of Antimicrobials
- Safety cohort (No Intervention): Cohort of patients with bacteremia due to carbapenem-resistant Acinetobacter baumannii and Pseudomonas aeruginosa, carbapenem-resistant enterobacteria, vancomycin-resistant Enterococcus faecium and methicillin-resistant Staphylococcus aureus occurred in participating hospitals from 2017 to 2021 will be collected.

INTERVENTIONS:
Behavioral: Non-impositive Program for Optimizing the Use of Antimicrobials — Quasi-experimental intervention through the development of a Program for Optimizing the Use of Antimicrobials in the participating hospitals. The intervention will consist of the development of a consensus guide on the use of new antibiotics, its dissemination in Andalusian hospitals and an audit on the prescription of new antibiotics.
  Arms: Intervention cohort

SUMMARY:
Quasi-experimental intervention multicenter trial of patients treated with new antibiotics (before-after study).

The study will be carried out in 14 hospitals of the Andalusian Public Health System with representation from all the provinces and has been designed in two phases:

1. A first phase in which an observational study of historical preintervention cohorts of patients who have received either empirical or targeted treatment with ceftaroline, tedizolid, dalbavancin, ceftazidime-avibactam, ceftolozane-tazobactam and isavuconazole from January 2016 to December 2019 will be developed. Case detection will be carried out by locating the antimicrobial prescriptions in the electronic prescribing systems and / or pharmaceutical management systems of each hospital. A set of epidemiological, clinical, microbiological and prognostic variables will be completed in each case.
2. A second phase or intervention period that will be applied to the cohort of patients treated with new antibiotics (intervention cohort) from January 2020 to June 2021. A quasi-experimental intervention study will be carried out through the development of a Program for Optimizing the use of Antibiotics (PROA) in Spanish, Antimicrobial Stewardship Program (ASP) in English, in the participating hospitals. It will consist in the development of a consensus document on the use of new antibiotics following a Delphi methodology, dissemination of the consensus document / guide among the participating hospitals and audit on the prescription of new antimicrobials after the implementation of the guide based on providing non-imposition advice and positive reinforcement to the prescriber. The recommendations will be consigned in a structured form, which will allow to evaluate the degree of follow-up of the recommendations. The audit will be performed on day 0-1 of the prescription.
3. Cohort of bacteremia due to multiresistant microorganisms ("safety" cohort): In order to evaluate the safety of the use of new antimicrobials against therapeutic alternatives in syndromes where they are potentially a preferred option and parallel to the two phases, episodes for bacteremia by carbapenem-resistant Acinetobacter baumannii and Pseudomonas aeruginosa, carbapenem-resistant enterobacteria, vancomycin-resistant Enterococcus faecium and methicillin-resistant Staphylococcus aureus occurred in participating hospitals from 2017 to 2021 will be collected.

ELIGIBILITY:
Pre-intervention cohort (historical):

Inclusion criteria:

* All patients treated with ceftaroline, tedizolid, dalbavancin, ceftazidime-avibactam, ceftolozane-tazobactam or isavuconazole.
* In a hospital or ambulatory regime.
* That they have received at least 1 dose of treatment of any of the antimicrobials mentioned, either as empirical or directed treatment.
* Adults (18 years).
* Between January 1, 2016 and December 31, 2019.

Exclusion criteria:

• There are no exclusion criteria except for age.

Intervention cohort:

Inclusion criteria:

* All patients treated with ceftaroline, tedizolid, dalbavancin, ceftazidime-avibactam, ceftolozane-tazobactam or isavuconazole.
* In a hospital or ambulatory regime.
* That they have received at least 1 dose of treatment of any of the antimicrobials mentioned, either as empirical or directed treatment.
* Adults (18 years).
* From January 1, 2020 to December 31, 2021.
* Since the publication and diffusion of the recommendation guide.

Exclusion criteria:

• There are no exclusion criteria except for age.

Safety cohort:

Inclusion criteria:

* All episodes of clinically significant bacteremia (that have received any treatment) produced by:
* Acinetobacter baumannii resistant or with intermediate susceptibility to any carbapenem.
* Pseudomonas aeruginosa resistant or with intermediate susceptibility to any carbapenem.
* Enterobacteria resistant or with intermediate susceptibility to any carbapenem.
* Vancomycin-resistant Enterococcus faecium.
* Methicillin-resistant Staphylococcus aureus.
* From January 1, 2017 to December 31, 2021.
* Adult patients (18 years old).

Exclusion criteria:

• There are no exclusion criteria except for age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Total antibiotic consumption | Yearly from date of intervention up to 24 months of follow-up
  Defined daily doses (DDD) of each antibiotic per 1000 stays

SECONDARY OUTCOMES:
Total cost per antimicrobial | Yearly from date of intervention up to 24 months of follow-up
  Total expense in euros of each antimicrobial per 1000 stays
Mortality rate | At 7, 14 and 30 days after the start of the treatment.
  Mortality from any cause at 7, 14 and 30 days after the start of the treatment.
Total length of hospital stay | Monthly from date of intervention up to 24 months of follow-up
  Duration of a single episode of hospitalization defined as the time between hospital admission and discharge measured in days. During this episode the patient has to be prescribed with one of the antibiotics included in the study.
Incidence of colitis due to Clostridium difficile. | Monthly from date of intervention up to 24 months of follow-up
  Clostridium difficile infection documented during treatment with any of the antibiotics described
Percentage of patients with infections by multiresistant microorganisms. Colonization during treatment by resistant microorganisms | Monthly from date of intervention up to 24 months of follow-up
  Percentage of patients with infections by multiresistant microorganisms in each cohort.
Percentage of patients colonized by multiresistant microorganisms | Monthly from date of intervention up to 24 months of follow-up
  Percentage of patients colonized by multiresistant microorganisms in each cohort after completion of treatment with antibiotic under study.
Re-admission rate | 90 days after the start of the antibiotic treatment.
  Re-admission of the patient in the hospital at 90 days after the start of the antibiotic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zaira Palacios Baena, Principal Investigator — University Hospital Virgen Macarena
Locations (14):
- Spain (14):
  - Hospital de Poniente-El Ejido, Almería
  - University Hospital Puerta del Mar, Cadiz
  - University Hospital Reina Sofía, Córdoba
  - Hospital Clínico Universitario San Cecilio, Granada
  - University Hospital Virgen de las Nieves, Granada
  - Área Hospitalaria Juan Ramón Jiménez, Huelva
  - Complejo Hospitalario de Jaén, Jaén
  - University Hospital de Jerez de la Frontera, Jerez de la Frontera
  - Hospital Regional Universitario de Málaga, Málaga
  - University Hospital Virgen de la Victoria, Málaga
  - Hospital de Puerto Real, Puerto Real
  - University Hospital Virgen de Valme, Seville
  - University Hospital Virgen del Rocío, Seville
  - University Hospital Virgen Macarena (Sevilla)., Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Versporten A, Zarb P, Caniaux I, Gros MF, Drapier N, Miller M, Jarlier V, Nathwani D, Goossens H; Global-PPS network. Antimicrobial consumption and resistance in adult hospital inpatients in 53 countries: results of an internet-based global point prevalence survey. Lancet Glob Health. 2018 Jun;6(6):e619-e629. doi: 10.1016/S2214-109X(18)30186-4. Epub 2018 Apr 23. PMID 29681513
- [Background] Rodriguez-Bano J, Cisneros JM, Cobos-Trigueros N, Fresco G, Navarro-San Francisco C, Gudiol C, Horcajada JP, Lopez-Cerero L, Martinez JA, Molina J, Montero M, Pano-Pardo JR, Pascual A, Pena C, Pintado V, Retamar P, Tomas M, Borges-Sa M, Garnacho-Montero J, Bou G; Study Group of Nosocomial Infections (GEIH) of the Spanish Society of Infectious Diseases, Infectious Diseases (SEIMC). Diagnosis and antimicrobial treatment of invasive infections due to multidrug-resistant Enterobacteriaceae. Guidelines of the Spanish Society of Infectious Diseases and Clinical Microbiology. Enferm Infecc Microbiol Clin. 2015 May;33(5):337.e1-337.e21. doi: 10.1016/j.eimc.2014.11.009. Epub 2015 Jan 15. PMID 25600218
- [Background] Lopez Cortes LE, Mujal Martinez A, Fernandez Martinez de Mandojana M, Martin N, Gil Bermejo M, Sola Aznar J, Villegas Bruguera E, Pelaez Cantero MJ, Retamar Gentil P, Delgado Vicente M, Gonzalez-Ramallo VJ, Ponce Gonzalez MA, Miron Rubio M, Gomez Rodriguez de Mendarozqueta MM, Goenaga Sanchez MA, Sanroma Mendizabal P, Delgado Mejia E, Pajaron Guerrero M; Sociedad Espanola de Enfermedades Infecciosas y Microbiologia Clinica (SEIMC), the Sociedad Espanola de Hospitalizacion a Domicilio (SEHAD) Group. Executive summary of outpatient parenteral antimicrobial therapy: Guidelines of the Spanish Society of Clinical Microbiology and Infectious Diseases and the Spanish Domiciliary Hospitalisation Society. Enferm Infecc Microbiol Clin (Engl Ed). 2019 Jun-Jul;37(6):405-409. doi: 10.1016/j.eimc.2018.03.012. Epub 2018 May 18. English, Spanish. PMID 29784453
- [Background] Tacconelli E, Carrara E, Savoldi A, Harbarth S, Mendelson M, Monnet DL, Pulcini C, Kahlmeter G, Kluytmans J, Carmeli Y, Ouellette M, Outterson K, Patel J, Cavaleri M, Cox EM, Houchens CR, Grayson ML, Hansen P, Singh N, Theuretzbacher U, Magrini N; WHO Pathogens Priority List Working Group. Discovery, research, and development of new antibiotics: the WHO priority list of antibiotic-resistant bacteria and tuberculosis. Lancet Infect Dis. 2018 Mar;18(3):318-327. doi: 10.1016/S1473-3099(17)30753-3. Epub 2017 Dec 21. PMID 29276051
- [Background] Plan estratégico y de acción para reducir el riesgo de selección y diseminación de la resistencia a los antibióticos http://www.resistenciaantibioticos.es/es/system/files/ content_images/plan_nacional_resistencia_antibioticos.pdf
- [Background] Rodriguez-Bano J, Pano-Pardo JR, Alvarez-Rocha L, Asensio A, Calbo E, Cercenado E, Cisneros JM, Cobo J, Delgado O, Garnacho-Montero J, Grau S, Horcajada JP, Hornero A, Murillas-Angoiti J, Oliver A, Padilla B, Pasquau J, Pujol M, Ruiz-Garbajosa P, San Juan R, Sierra R; GEIH-SEIMC; SEFH; SEMPSPH. [Programs for optimizing the use of antibiotics (PROA) in Spanish hospitals: GEIH-SEIMC, SEFH and SEMPSPH consensus document]. Farm Hosp. 2012 Jan-Feb;36(1):33.e1-30. doi: 10.1016/j.farma.2011.10.001. Epub 2011 Dec 1. Spanish. PMID 22137161
- [Background] Programa integral de prevención y control de las infecciones relacionadas con la asistencia sanitaria y uso apropiado de los antimicrobianos (PIRASOA). pirasoa.iavante.es/
- [Background] European Centre for Disease Prevention and Control. Rapid risk assessment: Carbapenem-resistant Enterobacteriaceae - first update 4 June 2018. Stockholm: ECDC; 2018. https://ecdc.europa.eu/sites/portal/files/documents/RRA-Enterobacteriaceae-Carbapenems-European-Union-countries.pdf
- [Background] Lopez-Cerero L, Egea P, Gracia-Ahufinger I, Gonzalez-Padilla M, Rodriguez-Lopez F, Rodriguez-Bano J, Pascual A. Characterisation of the first ongoing outbreak due to KPC-3-producing Klebsiella pneumoniae (ST512) in Spain. Int J Antimicrob Agents. 2014 Dec;44(6):538-40. doi: 10.1016/j.ijantimicag.2014.08.006. Epub 2014 Sep 26. PMID 25446907
- [Background] PIRASOA: actividad laboratorio de referencia. Accesible en: pirasoa.iavante.es/mod/resource/view.php?id=797
- [Background] Rodriguez-Bano J, Gutierrez-Gutierrez B, Machuca I, Pascual A. Treatment of Infections Caused by Extended-Spectrum-Beta-Lactamase-, AmpC-, and Carbapenemase-Producing Enterobacteriaceae. Clin Microbiol Rev. 2018 Feb 14;31(2):e00079-17. doi: 10.1128/CMR.00079-17. Print 2018 Apr. PMID 29444952
- [Background] Mensa J, Soriano A, Llinares P, Barberan J, Montejo M, Salavert M, Alvarez-Rocha L, Maseda E, Moreno A, Pasquau J, Gomez J, Parra J, Candel F, Azanza JR, Garcia JE, Marco F, Soy D, Grau S, Arias J, Fortun J, de Alarcon CA, Picazo J; Sociedad Espanola de Quimioterapia (SEQ); Sociedad Espanola de Medicina Interna (SEMI); GTIPO-Sociedad Espanola de Anestesiologia y Reanimacion. [Guidelines for antimicrobial treatment of the infection by Staphylococcus aureus]. Rev Esp Quimioter. 2013 Jan;26 Suppl 1:1-84. No abstract available. Spanish. PMID 23824510
- [Background] Spellberg B, Bonomo RA. Editorial Commentary: Ceftazidime-Avibactam and Carbapenem-Resistant Enterobacteriaceae: "We're Gonna Need a Bigger Boat". Clin Infect Dis. 2016 Dec 15;63(12):1619-1621. doi: 10.1093/cid/ciw639. Epub 2016 Sep 13. No abstract available. PMID 27624957
- [Background] Ficha técnica de ceftarolina. https://ec.europa.eu/health/documents/communityregister/2012/20120823123835/anx_123835_es.pdf
- [Background] Ficha técnica de tedizolid. http://www.ema.europa.eu/docs/es_ES/document_library /EPAR_-_Product_Information/human/002846/WC500184802.pdf
- [Background] Informa de posicionamiento terapéutico de dalbavancina. https://www.aemps.gob.es/medicamentosUsoHumano/informesPublicos/docs/IPTdalbavancina-Xydalba.pdf
- [Background] Ficha técnica de ceftazidima-avibactam. http://www.ema.europa.eu/docs/es_ES /document_library /EPAR_-_Product_Information/human/004027/WC500210234.pdf
- [Background] Ficha técnica de ceftolozano-tazobactam. https://ec.europa.eu/health/documents /communityregister/2015/20150918132786/anx_132786_es.pdf
- [Background] Ficha técnica de isavuconazol. https://ec.europa.eu/health/documents/community-register/2015/20151015132781/anx_132781_es.pdf.
- [Background] Cosimi RA, Beik N, Kubiak DW, Johnson JA. Ceftaroline for Severe Methicillin-Resistant Staphylococcus aureus Infections: A Systematic Review. Open Forum Infect Dis. 2017 May 2;4(2):ofx084. doi: 10.1093/ofid/ofx084. eCollection 2017 Spring. PMID 28702467
- [Background] Zasowski EJ, Trinh TD, Claeys KC, Casapao AM, Sabagha N, Lagnf AM, Klinker KP, Davis SL, Rybak MJ. Multicenter Observational Study of Ceftaroline Fosamil for Methicillin-Resistant Staphylococcus aureus Bloodstream Infections. Antimicrob Agents Chemother. 2017 Jan 24;61(2):e02015-16. doi: 10.1128/AAC.02015-16. Print 2017 Feb. PMID 27895012
- [Background] Si S, Durkin MJ, Mercier MM, Yarbrough ML, Liang SY. Successful Treatment of Prosthetic Joint Infection due to Vancomycin-resistant Enterococci with Tedizolid. Infect Dis Clin Pract (Baltim Md). 2017 Mar;25(2):105-107. doi: 10.1097/IPC.0000000000000469. PMID 28428726
- [Background] Nigo M, Luce AM, Arias CA. Long-term Use of Tedizolid as Suppressive Therapy for Recurrent Methicillin-Resistant Staphylococcus aureus Graft Infection. Clin Infect Dis. 2018 Jun 1;66(12):1975-1976. doi: 10.1093/cid/ciy041. No abstract available. PMID 29370350
- [Background] Tobudic S, Forstner C, Burgmann H, Lagler H, Ramharter M, Steininger C, Vossen MG, Winkler S, Thalhammer F. Dalbavancin as Primary and Sequential Treatment for Gram-Positive Infective Endocarditis: 2-Year Experience at the General Hospital of Vienna. Clin Infect Dis. 2018 Aug 16;67(5):795-798. doi: 10.1093/cid/ciy279. PMID 29659732
- [Background] Bouza E, Valerio M, Soriano A, Morata L, Carus EG, Rodriguez-Gonzalez C, Hidalgo-Tenorio MC, Plata A, Munoz P, Vena A; DALBUSE Study Group (Dalbavancina: Estudio de su uso clinico en Espana). Dalbavancin in the treatment of different gram-positive infections: a real-life experience. Int J Antimicrob Agents. 2018 Apr;51(4):571-577. doi: 10.1016/j.ijantimicag.2017.11.008. Epub 2017 Nov 24. PMID 29180276
- [Background] Iacovelli A, Spaziante M, Al Moghazi S, Giordano A, Ceccarelli G, Venditti M. A challenging case of carbapenemase-producing Klebsiella pneumoniae septic thrombophlebitis and right mural endocarditis successfully treated with ceftazidime/avibactam. Infection. 2018 Oct;46(5):721-724. doi: 10.1007/s15010-018-1166-9. Epub 2018 Jun 20. PMID 29926399
- [Background] Gofman N, To K, Whitman M, Garcia-Morales E. Successful treatment of ventriculitis caused by Pseudomonas aeruginosa and carbapenem-resistant Klebsiella pneumoniae with i.v. ceftazidime-avibactam and intrathecal amikacin. Am J Health Syst Pharm. 2018 Jul 1;75(13):953-957. doi: 10.2146/ajhp170632. PMID 29941534
- [Background] De Leon-Borras R, Alvarez-Cardona J, Vidal JA, Guiot HM. Ceftazidime/Avibactam for Refractory Bacteremia, Vertebral Diskitis/Osteomyelitis with Pre-Vertebral Abscess and Bilateral Psoas Pyomyositis Secondary to Klebsiella Pneumoniae Carbapenemase-Producing Bacteria (KPC). P R Health Sci J. 2018 Jun;37(2):128-131. PMID 29905925
- [Background] Dietl B, Sanchez I, Arcenillas P, Cuchi E, Gomez L, Gonzalez de Molina FJ, Boix-Palop L, Nicolas J, Calbo E. Ceftolozane/tazobactam in the treatment of osteomyelitis and skin and soft-tissue infections due to extensively drug-resistant Pseudomonas aeruginosa: clinical and microbiological outcomes. Int J Antimicrob Agents. 2018 Mar;51(3):498-502. doi: 10.1016/j.ijantimicag.2017.11.003. Epub 2017 Nov 20. PMID 29158144
- [Background] Vickery SB, McClain D, Wargo KA. Successful Use of Ceftolozane-Tazobactam to Treat a Pulmonary Exacerbation of Cystic Fibrosis Caused by Multidrug-Resistant Pseudomonas aeruginosa. Pharmacotherapy. 2016 Oct;36(10):e154-e159. doi: 10.1002/phar.1825. Epub 2016 Sep 1. PMID 27522066
- [Background] Plant AJ, Dunn A, Porter RJ. Ceftolozane-tazobactam resistance induced in vivo during the treatment of MDR Pseudomonas aeruginosa pneumonia. Expert Rev Anti Infect Ther. 2018 May;16(5):367-368. doi: 10.1080/14787210.2018.1473079. No abstract available. PMID 29727213
- [Background] Gaibani P, Campoli C, Lewis RE, Volpe SL, Scaltriti E, Giannella M, Pongolini S, Berlingeri A, Cristini F, Bartoletti M, Tedeschi S, Ambretti S. In vivo evolution of resistant subpopulations of KPC-producing Klebsiella pneumoniae during ceftazidime/avibactam treatment. J Antimicrob Chemother. 2018 Jun 1;73(6):1525-1529. doi: 10.1093/jac/dky082. PMID 29566151
- [Background] Davey P, Marwick CA, Scott CL, Charani E, McNeil K, Brown E, Gould IM, Ramsay CR, Michie S. Interventions to improve antibiotic prescribing practices for hospital inpatients. Cochrane Database Syst Rev. 2017 Feb 9;2(2):CD003543. doi: 10.1002/14651858.CD003543.pub4. PMID 28178770
- [Background] Diamond IR, Grant RC, Feldman BM, Pencharz PB, Ling SC, Moore AM, Wales PW. Defining consensus: a systematic review recommends methodologic criteria for reporting of Delphi studies. J Clin Epidemiol. 2014 Apr;67(4):401-9. doi: 10.1016/j.jclinepi.2013.12.002. PMID 24581294
- [Derived] Palacios-Baena ZR, Valiente de Santis L, Maldonado N, Rosso-Fernandez CM, Borreguero I, Herrero-Rodriguez C, Lopez-Cardenas S, Martinez-Marcos FJ, Martin-Aspas A, Jimenez-Aguilar P, Caston JJ, Anguita-Santos F, Ojeda-Burgos G, Aznarte-Padial MP, Praena-Segovia J, Corzo-Delgado JE, Esteban-Moreno MA, Rodriguez-Bano J, Retamar P. Quasiexperimental intervention study protocol to optimise the use of new antibiotics in Spain: the NEW_SAFE project. BMJ Open. 2020 Jul 31;10(7):e035460. doi: 10.1136/bmjopen-2019-035460. PMID 32737088